CLINICAL TRIAL: NCT02223494
Title: An Open-label, Long-term Safety Evaluation of Terbogrel in Patients With Primary Pulmonary Hypertension
Brief Title: Safety of Terbogrel in Patients With Primary Pulmonary Hypertension
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 528.21
Record Dates: First submitted 2014-08-21; First posted 2014-08-22 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Hypertension, Pulmonary
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — terbogrel

ARMS (1):
- Terbogrel (Experimental)
  Interventions: Drug: Terbogrel

INTERVENTIONS:
Drug: Terbogrel

SUMMARY:
Study to assess the safety of terbogrel during open-label, long-term treatment in medically stable or improving patients with primary pulmonary hypertension who have completed the 12-week, double-blind randomized trial of terbogrel (protocol 528.19)

ELIGIBILITY:
Inclusion Criteria:

Patients who

* completed the preceding primary pulmonary hypertension, double-blinded clinical trial of terbogrel (protocol 528.19)
* provide informed consent to participate in this trial
* are in a stable or improving medical condition, in the opinion of the investigator
* enter the study immediately upon their completion of the preceding double-blind Trial 528.19, or enter the study within one month of completing the preceding trial as long as their medical condition has remained stable or continues to improve in the interim

Exclusion Criteria:

* Development of an unstable medical condition during or following completion of the preceding clinical trial which, in the investigator's opinion, may be worsened by treatment with terbogrel
* Premature discontinuation of the preceding terbogrel clinical trial due to an adverse event or for any other reason
* Pregnant or nursing women, or women of childbearing potential (less than one year postmenopausal or not surgically sterilized) who are not using adequate methods of birth control

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 1998-10; Primary Completion 2000-03 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | up to 18 months
Number of patients with clinically significant findings in laboratory tests | up to 18 months
Number of patients with clinically significant changes in ECG | up to 18 months

SECONDARY OUTCOMES:
Change in patient status | baseline, up to 18 months
  change in New York Health Association (NYHA) class, need for treatment with Flolan or transplantation, death